CLINICAL TRIAL: NCT03569891
Title: Phase III, Open-label, Single-dose, Multi-center, Multinational Trial Investigating a Serotype 5 Adeno-associated Viral Vector Containing the Padua Variant of a Codon-optimized Human Factor IX Gene (AAV5-hFIXco-Padua, AMT-061) Administered to Adult Subjects With Severe or Moderately Severe Hemophilia B
Brief Title: HOPE-B: Trial of AMT-061 in Severe or Moderately Severe Hemophilia B Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CSL222_3001 (CT-AMT-061-02)
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Results first posted 2022-10-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Hemophilia B
Keywords: Gene therapy; FIX; factor IX; Bleeding; Viral vector; Padua; hemophilia; AAV (adeno-associated virus); serotype 5 AAV (adeno-associated virus); serotype 5
MeSH Terms: conditions — Hemophilia B; Hemorrhage; Hemophilia A | interventions — Factor IX

STUDY DESIGN:
Intervention Model Description: The reference therapy is prophylactic factor IX replacement therapy used during the lead-in phase prior to treatment with AAV5-hFIXco-Padua (AMT-061).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMT-061 (Experimental): Single infusion of AMT-061
  Subjects will receive a single infusion of AAV5-hFIXco-Padua (AMT- 061) at baseline. After study drug administration (post study drug), subjects will be monitored for tolerance to the study drug and detection of potential immediate AEs at the clinical trial site for a few hours after dosing.
  Interventions: Genetic: AAV5-hFIXco-Padua
- FIX replacement (Lead-in Period) (Active Comparator): During the lead-in phase, which lasted for a minimum of 26 weeks (i.e., ≥6 months), subjects recorded their use of FIX replacement therapy and bleeding episodes in their dedicated e-diary.
  Interventions: Biological: Factor IX (FIX)

INTERVENTIONS:
Genetic: AAV5-hFIXco-Padua — Single intravenous infusion of AAV5-hFIXco-Padua (AMT-061)
  Other Names: AMT-061; etranacogene dezaparvovec
  Arms: AMT-061
Biological: Factor IX (FIX) — During the lead-in phase, which lasted for a minimum of 26 weeks (i.e., ≥6 months), subjects recorded their use of FIX replacement therapy and bleeding episodes in their dedicated e-diary.
  Arms: FIX replacement (Lead-in Period)

SUMMARY:
This is an open-label, single-dose, multi-center, multinational trial to demonstrate the efficacy of AMT-061 and to further describe its safety profile.

The study drug is identified as AAV5-hFIXco-Padua (AMT- 061). AMT-061 is a recombinant adeno-associated viral vector of serotype 5 (AAV5) containing the Padua variant of a codon-optimized human FIX complementary deoxyribonucleic acid (cDNA) under the control of a liver-specific promoter. The pharmaceutical form of AMT-061 is a solution for intravenous infusion administered at a dose of 2 x 10^13 gc/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age ≥18 years
3. Subjects with congenital hemophilia B, classified as severe or moderately severe, and are currently on factor IX prophylaxis
4. >150 previous exposure days of treatment with factor IX protein

Exclusion Criteria:

1. History of factor IX inhibitors
2. Positive factor IX inhibitor test at screening
3. Select screening laboratory value >2 times upper limit of normal
4. Positive human immunodeficiency virus (HIV) test at screening, not controlled with anti-viral therapy
5. Active infection with hepatitis B or C virus at screening
6. History of Hepatitis B or C exposure, currently controlled by antiviral therapy at the end of the lead-in phase
7. Previous gene therapy treatment
8. Receipt of an experimental agent within 60 days prior to screening
9. Current participation or anticipated participation within one year after study drug administration in this trial in any other interventional clinical trial involving drugs or devices

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2025-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pipe, MD, Principal Investigator — University of Michigan
Locations (33):
- United States (19):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Los Angeles Orthopedic Hospital, Los Angeles, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - University of California, San Diego, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - Children's National Medical Center Hematology and Oncology, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Hemophilia Center of Western New York, Buffalo, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center & Medical School, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Washington Institute for Coagulation, Seattle, Washington
  - Bloodworks Northwest, Seattle, Washington
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital Leuven, Leuven
- Righospitalet, Copenhagen, Denmark
- Germany (2):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Klinikum der Johann Wolfgang Goethe Universitat, Frankfurt am Main
- National Coagulation Centre, St James's Hospital, Dublin, Ireland
- Netherlands (4):
  - Amsterdam UMC - Locatie AMC, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Van Creveldkliniek, Utrecht
- Center for Thrombosis and Hemostasis Skåne University Hospital Malmö, Malmo, Sweden
- United Kingdom (3):
  - The Cambridge Haemophilia and Thrombophilia Centre Camridge University Hospitals NHS Foundation Trust - Box 217 Addenbrooke's Hospital, Cambridge
  - The Royal London Hospital (Barts Health NHS Trust), London
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pipe SW, Miesbach W, Recht M, Leebeek FWG, Key NS, Castaman G, Lattimore S, Coppens M, Le Quellec S, Mahajan V, Gill S, Drelich D, Monahan PE; HOPE-B Study Group Investigators. Final Analysis of a Study of Etranacogene Dezaparvovec for Hemophilia B. N Engl J Med. 2026 Jan 29;394(5):463-474. doi: 10.1056/NEJMoa2514332. Epub 2025 Dec 7. PMID 41358585
- [Derived] O'Connell N, van der Valk P, Le Quellec S, Gomez E, Monahan PE, Crary SE, Coppens M, Lemons R, Castaman G, Klamroth R, Symington E, Quon DV, Kampmann P. Invasive procedures and surgery following etranacogene dezaparvovec gene therapy in people with hemophilia B. J Thromb Haemost. 2025 Jan;23(1):73-84. doi: 10.1016/j.jtha.2024.08.027. Epub 2024 Sep 26. PMID 39341368
- [Derived] Coppens M, Pipe SW, Miesbach W, Astermark J, Recht M, van der Valk P, Ewenstein B, Pinachyan K, Galante N, Le Quellec S, Monahan PE, Leebeek FWG; HOPE-B Investigators. Etranacogene dezaparvovec gene therapy for haemophilia B (HOPE-B): 24-month post-hoc efficacy and safety data from a single-arm, multicentre, phase 3 trial. Lancet Haematol. 2024 Apr;11(4):e265-e275. doi: 10.1016/S2352-3026(24)00006-1. Epub 2024 Mar 1. PMID 38437857
- [Derived] Pipe SW, Leebeek FWG, Recht M, Key NS, Castaman G, Miesbach W, Lattimore S, Peerlinck K, Van der Valk P, Coppens M, Kampmann P, Meijer K, O'Connell N, Pasi KJ, Hart DP, Kazmi R, Astermark J, Hermans CRJR, Klamroth R, Lemons R, Visweshwar N, von Drygalski A, Young G, Crary SE, Escobar M, Gomez E, Kruse-Jarres R, Quon DV, Symington E, Wang M, Wheeler AP, Gut R, Liu YP, Dolmetsch RE, Cooper DL, Li Y, Goldstein B, Monahan PE. Gene Therapy with Etranacogene Dezaparvovec for Hemophilia B. N Engl J Med. 2023 Feb 23;388(8):706-718. doi: 10.1056/NEJMoa2211644. PMID 36812434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an 18-month post-dose interim analysis due to the completion of the primary endpoint. The study will complete approximately 5 years after post-dose.
Pre-assignment Details: Sixty seven (67) participants were enrolled. Of those, 54 completed the Lead-in and were dosed with AMT-061.
Groups:
- Lead-in Safety Population: This is an 18-month post-dose interim analysis due to the completion of the primary endpoint. The study will complete approximately 5 years after post-dose.
  The Lead-in Safety Population consisted of all subjects who were enrolled into the lead-in phase.
  During the lead-in, which lasted for a minimum of 26 weeks (i.e., ≥6 months), subjects recorded their use of Factor IX (FIX) replacement therapy and bleeding episodes in their dedicated e-diary. AMT-061 was administered after the Lead-in Period.
Period: Lead-in
Arm/Group | Lead-in Safety Population
Started | 67
Completed | 54
Not Completed | 13
Not completed — Ineligible during lead-in | 8
Not completed — Withdrawal by Subject | 3
Not completed — Risks related to COVID-19 | 2
Period: AMT-061
Arm/Group | Lead-in Safety Population
Started | 54
Completed | 53
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: During the lead-in phase, which lasted for a minimum of 26 weeks (i.e., ≥6 months), subjects recorded their use of FIX replacement therapy and bleeding episodes in their dedicated e-diary. After the lead-in phase, subjects received a single-dose of AMT-061.
Arm/Group | Safety Population
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 56
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 50
  More than one race | 7
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  Netherlands | 13
  Sweden | 2
  Belgium | 6
  United States | 26
  Ireland | 3
  United Kingdom | 7
  Italy | 5
  Germany | 2
  Denmark | 3

OUTCOME MEASURES:

1. Primary Outcome: Annualized Bleeding Rate (ABR) for All Bleeding Episodes
Description: ABR was calculated as the ratio of the number of bleeds to the number of days in the time interval multiplied by 365.25.
Time Frame: Lead-in period and months 7-18 post-treatment of AMT-061
Population: Full Analysis Set (FAS) included all subjects who were enrolled, entered the lead-in phase, were dosed with AMT-061, and provided at least 1 efficacy endpoint assessment for any efficacy endpoint subsequent to AMT-061 dosing. Subjects who were Lead-in Discontinuers were not included in the FAS.
Measure: Mean (95% Confidence Interval); unit: bleeds/year/subject
Groups:
- FIX (Lead-in): During the lead-in phase, which lasted for a minimum of 26 weeks (i.e., ≥6 months), subjects recorded their use of FIX replacement therapy and bleeding episodes in their dedicated e-diary.
- AMT-061: Single infusion of AMT-061
  Subjects will receive a single infusion of AAV5-hFIXco-Padua (AMT- 061) at baseline after lead-in.
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
bleeds/year/subject | 4.19 [3.22 to 5.45] | 1.51 [0.81 to 2.82]

2. Secondary Outcome: Factor IX Activity Levels After AMT-061 Dosing
Time Frame: Baseline and 6,12, and 18 months after AMT-061 dosing
Population: FAS.
Measure: Mean (Standard Deviation); unit: Factor IX activity (%)
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 0 | 54
Factor IX activity (%)
  Baseline |  | 1.19 (0.39)
  6 months: number analyzed (Participants) | 0 | 51
  6 months |  | 38.95 (18.72)
  12 months: number analyzed (Participants) | 0 | 50
  12 months |  | 41.48 (21.71)
  18 months: number analyzed (Participants) | 0 | 50
  18 months |  | 36.90 (21.40)

3. Secondary Outcome: Annualized Exogenous Factor IX Consumption
Time Frame: Lead-in period and months 0-6, 7-12, and 13-18 after AMT-061 dosing
Population: FAS
Measure: Mean (Standard Deviation); unit: IU/year
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
IU/year
  Lead-in: number analyzed (Participants) | 54 | 0
  Lead-in | 257,338.8 (149,013.1) |
  Months 0-6: number analyzed (Participants) | 0 | 54
  Months 0-6 |  | 12,912.9 (37,093.1)
  Months 7-12: number analyzed (Participants) | 0 | 54
  Months 7-12 |  | 8399.1 (29,720.9)
  Months 13-18: number analyzed (Participants) | 0 | 54
  Months 13-18 |  | 8486.6 (28,770.2)

4. Secondary Outcome: Adjusted Annualized Infusion Rate of FIX Replacement Therapy
Time Frame: Lead-in period and months 7-18 after AMT-061 dosing
Population: FAS.
Measure: Mean (95% Confidence Interval); unit: Infusions/year
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
Infusions/year
  Lead-in: number analyzed (Participants) | 54 | 0
  Lead-in | 72.49 [63.52 to 82.71] |
  Months 7-18: number analyzed (Participants) | 0 | 54
  Months 7-18 |  | 2.53 [0.92 to 6.96]

5. Secondary Outcome: Percent of Subjects Who Discontinued FIX Prophylaxis and Remained Free of Routine FIX Prophylaxis After AMT-061 Dosing
Time Frame: Months 7-18 after AMT-061 dosing
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | AMT-061
Number analyzed (Participants) | 54
percentage of participants | 96.3

6. Secondary Outcome: Percentage of Subjects With Trough FIX Activity <12% of Normal
Time Frame: Lead-in and 3, 12, and 18 months after AMT-061 dosing
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
percentage of participants
  Lead-in: number analyzed (Participants) | 54 | 0
  Lead-in | 79.6 |
  3 months: number analyzed (Participants) | 0 | 51
  3 months |  | 7.8
  12 months: number analyzed (Participants) | 0 | 50
  12 months |  | 8.0
  18 months: number analyzed (Participants) | 0 | 50
  18 months |  | 6.0

7. Secondary Outcome: ABR for FIX-treated Bleeding Episodes
Time Frame: Lead-in and Months 7-18 after AMT-061 dosing
Population: FAS
Measure: Mean (95% Confidence Interval); unit: bleeds/year/subject
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
bleeds/year/subject | 3.65 [2.82 to 4.74] | 0.84 [0.41 to 1.73]

8. Secondary Outcome: Number of Spontaneous Bleeding Episodes
Time Frame: Lead-in period and months 7-18 after AMT-061 dosing
Population: FAS
Measure: Number; unit: Number of bleeds
Groups:
- AMT-061: Single infusion of AMT-061
  Subjects will receive a single infusion of AAV5-hFIXco-Padua (AMT- 061) at baseline after lead-in .
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
Number of bleeds
  Lead-in: number analyzed (Participants) | 54 | 0
  Lead-in | 50 |
  Months 7-18: number analyzed (Participants) | 0 | 54
  Months 7-18 |  | 14

9. Secondary Outcome: Number of Joint Bleeding Episodes
Time Frame: Lead-in period and months 7-18 after AMT-061 dosing
Population: FAS
Measure: Number; unit: Number of bleeds
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
Number of bleeds
  Lead-in: number analyzed (Participants) | 54 | 0
  Lead-in | 77 |
  Months 7-18: number analyzed (Participants) | 0 | 54
  Months 7-18 |  | 19

10. Secondary Outcome: Mean FIX Activity (%) in Subjects With Pre-Existing Neutralizing Antibodies to AAV5 After AMT-061 Dosing
Time Frame: Baseline and 6,12, and 18 months after AMT-061 dosing
Population: FAS
Measure: Mean (Standard Deviation); unit: Factor IX activity (%)
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 0 | 21
Factor IX activity (%)
  Baseline |  | 1.24 (0.44)
  6 months: number analyzed (Participants) | 0 | 18
  6 months |  | 35.91 (19.02)
  12 months: number analyzed (Participants) | 0 | 18
  12 months |  | 35.54 (17.84)
  18 months: number analyzed (Participants) | 0 | 17
  18 months |  | 31.14 (13.75)

11. Secondary Outcome: Mean FIX Activity (%) in Subjects Without Pre-Existing Neutralizing Antibodies to AAV5 After AMT-061 Dosing
Time Frame: Baseline and 6,12, and 18 months after AMT-061 dosing
Population: FAS
Measure: Mean (Standard Deviation); unit: Factor IX activity (%)
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 0 | 33
Factor IX activity (%)
  Baseline |  | 1.15 (0.36)
  6 months |  | 40.61 (18.64)
  12 months: number analyzed (Participants) | 0 | 32
  12 months |  | 44.82 (23.21)
  18 months |  | 39.87 (24.08)

12. Secondary Outcome: Number of New Target Joints and the Number of New Target Joints Resolved.
Description: A target joint was defined as 3 or more spontaneous bleeding episodes into a single joint within a consecutive 6-month period prior to the dosing visit and which was not resolved by the time of dosing. An identified target joint with ≤2 spontaneous bleeding episodes within a consecutive 12-month period was considered resolved.
Time Frame: Up to 18 months after AT-061 dosing
Population: FAS
Measure: Number; unit: Joints
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 0 | 54
Joints
  New target joints |  | 1
  New target joints resolved |  | 0

13. Secondary Outcome: Percent of Participants With Zero Bleeding Episodes During the 52 Weeks Following Stable FIX Expression (6 to 18 Months) After AMT-061 Dosing
Time Frame: Lead-in period and months 7-18 post-treatment of AMT-061
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
percentage of participants | 25.9 | 63.0

14. Secondary Outcome: International Physical Activity Questionnaire (iPAQ) Overall Score
Description: The iPAQ was designed to provide an evaluation of daily physical activities in metabolic equivalent of task (MET) minutes/week. To calculate MET minutes a week multiply the MET value given (walking = 3.3, moderate activity = 4, vigorous activity = 8) by the minutes the activity was carried out and again by the number of days that that activity was undertaken. A higher score is considered to be more favorable.
Time Frame: Lead-in period and up to 12 months after AT-01 dosing
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: MET minutes/week
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
MET minutes/week | 4548.1 (512.38) | 3826.9 (480.44)

15. Secondary Outcome: EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) VAS Overall Score
Description: The EQ-5D-5L descriptive system of health-related QoL states consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The EQ-5D-5L VAS overall score ranges from 0 to 100. A higher score is considered to be more favorable.
Time Frame: Lead-in period and up to 12 months after AMT-061 dosing
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | FIX (Lead-in) | AMT-061
Number analyzed (Participants) | 54 | 54
score on a scale | 80.9 (2.20) | 81.0 (2.15)

16. Secondary Outcome: Number of Adverse Events
Description: Follow up and assess any adverse events reported for safety
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2026-03

ADVERSE EVENTS:
Time Frame: Up to 2 years per subject (up to 6 months Lead-in and up to an additional 18 months post-dose)
Description: This is an 18-month post-dose interim analysis due to the completion of the primary endpoint. The study will complete approximately 5 years after post-dose.
  The Safety Population consisted of all subjects who were enrolled in either the Lead-in Safety Population (consisted of all subjects who were enrolled into the lead-in phase) or the Post-treatment Safety Population (consisted of all subjects who received AMT-061, irrespective of any protocol deviations).
Groups:
- Lead-In (Including Discontinuers); Lead-In (Not Including Discontinuers): During the lead-in phase, which lasted for a minimum of 26 weeks (i.e., ≥6 months), subjects recorded their use of FIX replacement therapy and bleeding episodes in their dedicated e-diary.
- AMT-061: Single infusion of AMT-061 after lead-in.
Arm/Group | Lead-In (Including Discontinuers) | Lead-In (Not Including Discontinuers) | AMT-061
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/54 | 1/54
Serious Adverse Events (participants affected / at risk) | 5/67 | 4/54 | 13/54
Other Adverse Events (participants affected / at risk) | 27/67 | 24/54 | 53/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-In (Including Discontinuers) (N=67) | Lead-In (Not Including Discontinuers) (N=54) | AMT-061 (N=54)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Complication Associated With Device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead-In (Including Discontinuers) (N=67) | Lead-In (Not Including Discontinuers) (N=54) | AMT-061 (N=54)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 18 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 7 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 14 (16)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 7 (11)
Pain (General disorders) | 2 (2) | 1 (1) | 4 (4)
Malaise (General disorders) | 0 (0) | 0 (0) | 5 (7)
Chest pain (General disorders) | 0 (0) | 0 (0) | 4 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 3 (4)
Nasopharyngitis (Infections and infestations) | 8 (8) | 8 (8) | 15 (20)
Cystitis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (6)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (7)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 16 (31)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 11 (12)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 8 (10)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 7 (8)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 4 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 4 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 3 (3)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 4 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (4)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
This is an 18-month post-dose interim analysis due to the completion of the primary endpoint. The study will complete approximately 5 years after post-dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT03569891/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03569891/SAP_001.pdf